CLINICAL TRIAL: NCT06780722
Title: Study of the Occurrence of Cardiocirculatory Arrest as a Function of the Level of Hypoxemia During a Maastricht 3 Procedure. Prospective Observational Multicenter Study
Brief Title: Study of the Occurrence of Cardiocirculatory Arrest as a Function of the Level of Hypoxemia During a Maastricht 3 Procedure
Acronym: HEPHAISTOS
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0498
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest; Reanimation
MeSH Terms: conditions — Heart Arrest | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling — * The first sample is taken at the start of the therapeutic stop.
  * The second sample is taken when the mean arterial pressure drops to 45mmHg.
  * The third sample is taken when circulatory arrest occurs.
  * The fourth sample is taken at the start of extracorporeal circulation. These four samples will be destroyed at the end of the study.

SUMMARY:
Evaluation of the level of hypoxemia during the occurrence of cardiocirculatory arrest during a Maastricht III organ donation procedure.

DETAILED DESCRIPTION:
Evaluation of the level of hypoxemia during the occurrence of cardiocirculatory arrest during a Maastricht III organ donation procedure.

ELIGIBILITY:
FOR THE DONORS :

Inclusion Criteria :

* Patient over 18 years of age
* Organ donation procedure initiated in accordance with the legislation and procedures in force in France for the Maastricht III category
* No opposition formulated by the relative to the patient's participation in the study

Exclusion Criteria :

* Patient registered on the national register of refusals or living refusal of donation
* Pregnant or breast-feeding women
* Patients under guardianship, curatorship or legal protection
* Medical contraindication to organ donation according to the recommendations of the Agence de Biomédecine currently in force in France

FOR THE RECEIVER

Inclusion Criteria :

* No opposition to the collection of data concerning him/her
* Patient over 18 at pre-transplant consultation
* Patient who has received an organ from a donor participating in the HEPHAISTOS protocol

Exclusion Criteria :

- Patients under guardianship, curatorship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who may be candidates for an organ donation procedure in the event of death in intensive care following the implementation of a procedure to discontinue active therapies.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2027-06-19 (Estimated)

PRIMARY OUTCOMES:
PaO2 level | 24 hours
  PaO2 level and its 95% confidence interval in the event of circulatory cardiac arrest, defined as no electrical activity and a pulse pressure below 5 mmHg, during a Maastricht III procedure.

SECONDARY OUTCOMES:
Spo2 Level | 24 hours
  Define the level of Spo2 (and its 95% confidence interval) at the time of cardiocirculatory arrest during a Maastricht III procedure.
Time between occurrence of first episode of pulsed oxygen saturation below 95% and onset of cardiocirculatory arrest | 24 hours
  Define the time (and its 95% confidence interval) between the occurrence of the first first episode of pulsed oxygen saturation below 95% and the onset of cardio-circulatory arrest defined by absence of electrical activity and pulsed pressure below 5 mmHg.
Correlation between the rate of delayed recovery of renal function in the recipient and the presence of hypoxemia at the time of cardiocirculatory arrest in the donor. | 7 days
  Delayed recovery of renal function will be confirmed if the recipient undergoes dialysis within the first 7 days after transplantation. Hypoxemia is defined as a PaO2 less than or equal to the median value.

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU ANGERS - Réanimation médicale, Angers
  - CHU ANGERS - Urgences - Coordination Prélèvements, Angers
  - CH ANNECY GENEVOIS - Réanimation médicale - Coordination Prélèvements multi-organes, Annecy
  - CH AVIGNON - CH Henri Duffaut - Réanimation polyvalente, Avignon
  - CHD Vendée - Les Oudairies - Médecine Intensive Réanimation -Coordination Prélèvements multi-organes, La Roche-sur-Yon
  - CHD Vendée - Les Oudairies - Médecine Intensive Réanimation, La Roche-sur-Yon
  - CHU LILLE - Hôpital Roger Salengro - Coordination prélèvements multi-organes, Lille
  - CHU LILLE - Hôpital Roger Salengro - Médecine Intensive Réanimation, Lille
  - CHU NANTES +- Médecine Intensive Réanimation, Nantes
  - CHU Nantes - Coordination prélèvement multi organes, Nantes
  - CHRU ORLEANS -Médecine Intensive Réanimation - Coordination Prélèvements multi-organes, Orléans
  - APHP Hôpital COCHIN - Coordination Prélèvements d'Organes et Tissus, Paris
  - APHP Hôpital COCHIN - Médecine Intensive Réanimation, Paris
  - CH PERIGUEUX - Réanimation - Coordination Prélèvements Organes et Tissus, Périgueux
  - CHU POITIERS - Anesthésie Réanimation - Coordination Prélèvements multi-organes, Poitiers
  - CHU RENNES - CHU Pontchaillou - Réanimation médicale, Rennes
  - CHRU TOURS - Hôpital Bretonneau - Coordination Prélèvements multi-organes, Tours
  - CHRU TOURS - Hôpital Bretonneau - Médecine Intensive Réanimation, Tours
  - CHBA Vannes-Auray - Réanimation Polyvalente, Vannes